CLINICAL TRIAL: NCT04784455
Title: Multicentre Study of Nomacopan (rVA576) in Paediatric Haematopoietic Stem-Cell Transplant Associated Thrombotic Microangiopathy
Brief Title: Nomacopan (rVA576) in Transplant Associated Thrombotic Microangiopathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The early termination of this study is a business decision following a portfolio reprioritization plan. The decision is not related to any Efficacy, Safety or Clinical concerns regarding Nomacopan/rVA576
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK901
Record Dates: First submitted 2020-11-19; First posted 2021-03-05 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Thrombotic Microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Intervention Model Description: Open-label, uncontrolled, multi-centre two-part study. Part A: dose algorithm, safety and efficacy Part B: safety and efficacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nomacopan (rVA576) (Experimental): The study population will consist of paediatric patients who have undergone allogeneic or autologous haematopoietic stem cell transplantation (HSCT) and develop transplant-associated thrombotic microangiopathy (HSCT-TMA) within a year of HSCT
  Interventions: Drug: nomacopan (rVA576)

INTERVENTIONS:
Drug: nomacopan (rVA576) — The study population will consist of paediatric patients who have undergone allogeneic or autologous HSCT and develop HSCT-TMA within a year of HSCT

SUMMARY:
Multicentre Study of nomacopan in Paediatric Haematopoietic Stem-Cell Transplant Associated Thrombotic Microangiopathy

DETAILED DESCRIPTION:
This is an open-label, multi-centre study of two-parts, Part A and B, includes 24 weeks of treatment, safety follow up after 30 days.

Part A: dose algorithm, safety and efficacy

Part B: safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 0.5 and < 18 years at the time of diagnosis of TMA.
2. Undergone allogeneic or autologous HSCT.
3. TMA diagnosis within a year of their allogeneic or autologous HSCT.
4. Clinical or histological diagnosis of TMA
5. Provision of written informed consent.
6. Provision of informed assent

Exclusion Criteria:

1. Patients weighing less than 5 kg.
2. Patients with a positive direct Coombs' test.
3. Patients who do not receive nomacopan within 21 days of the initial diagnosis of TMA.
4. Patients having an active systemic or organ system bacterial or fungal infection or progressive severe infection at the time of diagnosis of TMA
5. Grade 4 Acute graft-versus-host disease (GVHD)
6. Received eculizumab or any other complement blocker therapy at any time.
7. Known hypersensitivity to the active ingredient or excipients

If an enrolled patient has a positive ADAMTS13 test (<10%) returned from their screening assessment, the patient should be withdrawn from the study

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Children's Hospital, Palo Alto, California
  - Duke University Medical Center, Children's Health Center, Durham, North Carolina
  - Children's Hospitall of Philadelphia, Philadelphia, Pennsylvania
- Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Poland
- United Kingdom (4):
  - The Royal Marsden NHS Foundation Trust, London
  - St. Georges University Hospital, London
  - Great Ormond Street Hospital (GOSH), London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consists of paediatric patients who have undergone allogeneic or autologous haematopoietic stem cell transplantation (HSCT) and developed haematopoietic stem cell transplant associated thrombotic microangiopathy (HSCT-TMA) within a year of HSCT
Groups:
- Nomacopan: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
Period: Overall Study
Arm/Group | Nomacopan
Started | 10
Completed | 6
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Nomacopan
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  ≥ 0.5 to < 2 years | 1
  ≥ 2 to < 9 years | 3
  ≥ 9 to < 18 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants NOT Requiring a Red Blood Bell Transfusion (Transfusion Independence) for 28 Days or More OR Number of Participants With a Urine Protein Creatinine Ratio Value of ≤ 2 mg/mg Maintained for 28 Days or More.
Description: Red blood cell transfusion independence for ≥28 days immediately prior to any scheduled clinical visit up to Week 24 or Urine protein creatinine ratio ≤ 2 mg/mg maintained over ≥ 28 days immediately prior to any scheduled clinical visit up to week 24
  Transfusion independence is defined as no RBC transfusion attributable to, or required to manage, thrombotic microangiopathy (TMA). Transfusions required for causes other than TMA will not be considered within the evaluation of the efficacy endpoints.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nomacopan
Number analyzed (Participants) | 10
Participants
  RBC transfusion independent for ≥ 28 days | 2
  Urine protein creatinine ratio (UPCR) ≤ 2 mg/mg for ≥ 28 days | 4

2. Secondary Outcome: Number of Participants With a Normalised sC5b-9 Value (Where sC5b-9 is the Same Value as the Upper Limit of Normal or Less)
Description: Plasma sC5b-9 ≤ upper limit of normal (ULN)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nomacopan
Number analyzed (Participants) | 10
Participants | 10

3. Secondary Outcome: Number of Participants With a Normalised Lactate Dehydrogenase (LDH) Value (Where LDH is the Same Value as the Upper Limit of Normal or Less)
Description: Lactate dehydrogenase (LDH) ≤ULN
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nomacopan
Number analyzed (Participants) | 10
Participants | 2

4. Secondary Outcome: Normalisation of Lab Parameters
Description: Number of participants with a normalised haptoglobin value (where haptoglobin is within the normal ranges)
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nomacopan
Number analyzed (Participants) | 10
Participants | 4

5. Secondary Outcome: Number of Participants Not Requiring a Platelet Transfusion (Transfusion Independence) for 28 Days or More.
Description: Transfusion independence is defined as no platelet transfusion attributable to, or required to manage, thrombotic microangiopathy (TMA). Transfusions required for causes other than TMA will not be considered within the evaluation of the efficacy endpoints.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Nomacopan: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
Arm/Group | Nomacopan
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: Duration of the study (Maximum of 2 year follow-up)
Description: An ablating dose was given on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1.
  One patient was administered the 1.7 mg/kg ablation dose, 3 patients received the 1.3 mg/kg ablation dose and 6 patients received the 1.0 mg/kg ablation dose.
  There were three maintenance dose levels - 0.3 mg/kg, 0.45 mg/kg and 0.60 mg/kg.
  All ten patients started on 0.3 mg/kg. Three patients had a dose escalation to 0.45mg/kg. No patient were dose escalated to 0.60 mg/kg.
Groups:
- Nomacopan - 1.7 mg/kg: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  One patient received the ablating dose of 1.7mg/kg.
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
- Nomacopan - 1.3 mg/kg: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  Three patients received the ablating dose of 1.7mg/kg.
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
- Nomacopan - 1.0 mg/kg: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  Six patients received the ablating dose of 1.7mg/kg.
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
- Nomacopan - 0.30 mg/kg: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
  10 patient received the starting dose of 0.30 mg/kg
- Nomacopan - 0.45 mg/kg: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
  Of the 10 enrolled patients, 3 patients had a dose increase to 0.45 mg/kg
- Nomacopan - 0.60 mg/kg: The trial was a 24-week open-label, non-comparative study in paediatric patients with HSCT-TMA.
  Patients will be given an ablating dose on Day 1, 12 hours apart which was determined by the child's age and weight on Day 1:
  Ablating Dose:
  * 0.5 to < 2 years =1.7 mg/kg
  * 2 to < 9 years =1.3 mg/kg
  * 9 to < 18 years =1.0 mg/kg
  For children in the youngest two cohorts (≥ 0.5 to < 2 years, and ≥ 2 to < 9 years), the dose was re-calculated at the week 8 and week 16 visits using the child's new weight measured at that visit.
  The starting maintenance dose, administered 12 hours apart, from Day 2 until the end of treatment was 0.30 mg/kg for all 3 age groups.
  If required, from pre-dose Day 7 onwards, a dose escalation was permitted if the CH50 results were > 10 U Eq/mL and/or the unbound nomacopan in serum was < 55 ng/mL.
  Two dose escalations were permitted - an increase from the maintenance dose of 0.30 mg/kg to 0.45 mg/kg with a further increase to 0.60 mg/kg if required. Dose increases were preceded by an ablating dose as determined by age as per Day 1.
  No patients had a dose increase to 0.60 mg/kg
Arm/Group | Nomacopan - 1.7 mg/kg | Nomacopan - 1.3 mg/kg | Nomacopan - 1.0 mg/kg | Nomacopan - 0.30 mg/kg | Nomacopan - 0.45 mg/kg | Nomacopan - 0.60 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/6 | 4/10 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/6 | 6/10 | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 1/6 | 7/10 | 2/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nomacopan - 1.7 mg/kg (N=1) | Nomacopan - 1.3 mg/kg (N=3) | Nomacopan - 1.0 mg/kg (N=6) | Nomacopan - 0.30 mg/kg (N=10) | Nomacopan - 0.45 mg/kg (N=3) | Nomacopan - 0.60 mg/kg (N=0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nomacopan - 1.7 mg/kg (N=1) | Nomacopan - 1.3 mg/kg (N=3) | Nomacopan - 1.0 mg/kg (N=6) | Nomacopan - 0.30 mg/kg (N=10) | Nomacopan - 0.45 mg/kg (N=3) | Nomacopan - 0.60 mg/kg (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (24) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (16) | 1 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (17) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (16) | 1 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 1 (3) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04784455/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04784455/SAP_001.pdf